CLINICAL TRIAL: NCT00245466
Title: An Open-Label, Multi-Centre, Extension Study Investigating the Long-Term Safety and Tolerability of Repeated Doses of Degarelix in Prostate Cancer Patients.
Brief Title: Study Investigating the Long-Term Safety and Tolerability of Repeated Doses of Degarelix in Prostate Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The maintenance doses were too low to maintain testosterone suppression
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS02A
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Results first posted 2009-06-11 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen ablation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Degarelix 80/80 + 40 (Experimental): In the main study (FE200486 CS02; NCT00819247) loading doses of degarelix 80 mg were given on Days 0 and 3. Maintenance doses of 40 mg were given on days 28, 56, 84, 112 and 140. In the extension study (FE200486 CS02A) the same maintenance dose of degarelix was given once every 4 weeks.
  Interventions: Drug: Degarelix
- Degarelix 40/40 + 40 (Experimental): In the main study (FE200486 CS02; NCT00819247) loading doses of degarelix 40 mg were given on Days 0 and 3. Maintenance doses of 40 mg were given on days 28, 56, 84, 112 and 140. In the extension study (FE200486 CS02A) the same maintenance dose of degarelix was given once every 4 weeks.
  Interventions: Drug: Degarelix
- Degarelix 80 + 20 (Experimental): In the main study (FE200486 CS02; NCT00819247) one loading dose of degarelix 80 mg was given on Days 0. Maintenance doses of 20 mg were given on days 28, 56, 84, 112 and 140. In the extension study (FE200486 CS02A) the same maintenance dose of degarelix was given once every 4 weeks.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Given as a subcutaneous injection once every 4 weeks.
  Other Names: FE200486
  Arms: Degarelix 80/80 + 40
Drug: Degarelix — Given as a subcutaneous injection once every 4 weeks.
  Other Names: FE200486
  Arms: Degarelix 40/40 + 40
Drug: Degarelix — Given as a subcutaneous injection once every 4 weeks.
  Other Names: FE200486
  Arms: Degarelix 80 + 20

SUMMARY:
To investigate the long-term safety and tolerability of repeated doses of degarelix to prostate cancer patients

DETAILED DESCRIPTION:
Degarelix was not FDA regulated at the time of the trial. After completion of the trial degarelix has been approved by the FDA and is thus an FDA regulated intervention (FDA regulated intervention is therefore ticked "YES").

The data include participants from both the main study (FE200486 CS02; NCT00819247) and the extension study FE200486 CS02A.

ELIGIBILITY:
Inclusion Criteria:

* Has completed study treatment in study FE200486 CS02.
* Has completed visit 16 in study FE200486 CS02.
* Has not met any withdrawal criteria up to and including visit 15 in FE200486 CS02

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2001-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who responded to degarelix in FE200486 CS02 (NCT00819247) were eligible to enroll into this extension study with the intention of continuing treatment until degarelix became commercially available in the UK or until the study was discontinued.
Groups:
- Degarelix 80/80 + 40: In the main study (FE200486 CS02) loading doses of degarelix 80 mg were given on Days 0 and 3. Maintenance doses of 40 mg were given on days 28, 56, 84, 112 and 140. In the extension study (FE200486 CS02A) the same maintenance dose of degarelix was given once every 4 weeks.
- Degarelix 40/40 + 40: In the main study (FE200486 CS02) loading doses of degarelix 40 mg were given on Days 0 and 3. Maintenance doses of 40 mg were given on days 28, 56, 84, 112 and 140. In the extension study (FE200486 CS02A) the same maintenance dose of degarelix was given once every 4 weeks.
- Degarelix 80 + 20: In the main study (FE200486 CS02) one loading dose of degarelix 80 mg was given on Days 0. Maintenance doses of 20 mg were given on days 28, 56, 84, 112 and 140. In the extension study (FE200486 CS02A) the same maintenance dose of degarelix was given once every 4 weeks.
Period: Overall Study
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Started | 43 | 46 | 40
Started FE200486 CS02A | 32 | 30 | 26
Completed | 7 (Defined as those participants ongoing when the extension study was terminated) | 2 | 3
Not Completed | 36 | 44 | 37
Not completed — Adverse Event | 2 | 8 | 4
Not completed — Low prostate specific antigen suppr | 16 | 14 | 5
Not completed — Insufficient testosterone suppr | 12 | 12 | 21
Not completed — Insufficient PSA and testosterone suppr | 0 | 0 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Disease progression | 0 | 3 | 1
Not completed — Protocol Violation | 1 | 2 | 2
Not completed — Death | 0 | 2 | 0
Not completed — Administrative reasons | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20 | Total
Number analyzed (Participants) | 43 | 46 | 40 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 7 | 18
  >=65 years | 37 | 41 | 33 | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 72.4 (6.60) | 73.7 (7.22) | 71.8 (7.08) | 72.7 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 43 | 46 | 40 | 129
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 1 | 3 | 1 | 5
  White | 42 | 43 | 37 | 122
  Indian | 0 | 0 | 1 | 1
  Afro-Carribean | 0 | 0 | 1 | 1
Gleason score [Number; unit: participants] — The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  participants
    Unknown | 1 | 1 | 1 | 3
    2-4 | 3 | 4 | 2 | 9
    5-6 | 11 | 7 | 11 | 29
    7-10 | 28 | 34 | 26 | 88
Number of Participants With Curative Intent [Number; unit: participants] — A curative intent of Yes refers to participants who have been castrated via radical prostatectomy or radiotherapy.
  participants
    Yes | 0 | 2 | 1 | 3
    No | 43 | 44 | 39 | 126
Number of Participants at Each Stage of Prostate Cancer [Number; unit: participants] — Prostate cancer stage was classified to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor.
  participants
    Localized | 8 | 9 | 5 | 22
    Locally advanced | 21 | 21 | 18 | 60
    Metastatic | 11 | 14 | 17 | 42
    Not classifiable | 3 | 2 | 0 | 5
Body mass index [Mean (Standard Deviation); unit: kilogram per square meter] — Body mass index is a measure of body fat based on height and weight.
  kilogram per square meter | 26.6 (4.15) | 26.6 (4.06) | 25.9 (3.93) | 26.4 (3.93)
Serum testosterone levels [Median (Inter-Quartile Range); unit: nanogram per milliliter] | 3.74 [3.08 to 4.94] | 4.11 [3.32 to 5.73] | 4.70 [3.54 to 5.77] | 3.98 [3.21 to 5.53]
Weight [Mean (Standard Deviation); unit: kilogram] | 77.6 (11.4) | 78.5 (14.2) | 76.3 (9.78) | 77.5 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Liver Function Tests
Description: The figures present the number of participants who had abnormal (defined as above upper limit of normal range (ULN)) alanine aminotransferase (ALT) levels, aspartate aminotransferase levels, and bilirubin levels plus the number of participants who had ALT increases >3x ULN and ALT increases >3x ULN with concurrently increased bilirubin >1.5 ULN.
Time Frame: 3 years
Population: The data include patients from both the main study (FE200486 CS02) and the extension study FE200486 CS02A.
Measure: Number; unit: participants
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Number analyzed (Participants) | 43 | 46 | 40
participants
  Abnormal alanine aminotransferase (ALAT) | 18 | 16 | 16
  Abnormal aspartate aminotransferase | 23 | 22 | 17
  Abnormal bilirubin | 3 | 4 | 5
  ALAT >3x ULN | 2 | 2 | 1
  ALAT >3x ULN, bilirubin >1.5x ULN | 0 | 0 | 1

2. Primary Outcome: Participants With Markedly Abnormal Change in Vital Signs and Body Weight
Description: Vital signs and body weight included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight at the end of trial as compared to baseline. The table presents the number of patients in each group with normal baseline and markedly abnormal value post-baseline.
Time Frame: 3 years
Population: These data include patients from the main study (FE200486 CS02) and the extension study (FE200486 CS02A).
Measure: Number; unit: participants
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Number analyzed (Participants) | 43 | 46 | 40
participants
  Diastolic blood pressure <=50 and decrease >=15 | 1 | 0 | 2
  Diastolic blood pressure >=105 and increase >=15 | 0 | 2 | 0
  Systolic blood pressure <=90 and decrease >=20 | 0 | 0 | 0
  Systolic blood pressure >=180 and increase >=20 | 8 | 7 | 1
  Heart rate <=50 and decrease >=15 | 0 | 1 | 2
  Heart rate >=120 and increase >=15 | 0 | 0 | 0
  Body weight decrease of >=7 percent | 5 | 4 | 5
  Body weight increase of >=7 percent | 17 | 14 | 15

3. Secondary Outcome: Serum Levels of Testosterone After 1, 2, and 3 Years
Time Frame: 3 years
Measure: Median (Full Range); unit: nanogram per milliliter
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Number analyzed (Participants) | 43 | 46 | 40
nanogram per milliliter
  1 year (n=25,17,14) | 0.120 [0.025 to 0.345] | 0.086 [0.025 to 0.372] | 0.170 [0.025 to 0.680]
  2 years (n=16,9,8) | 0.143 [0.025 to 0.805] | 0.133 [0.025 to 0.557] | 0.305 [0.064 to 0.454]
  3 years (n=8,5,6) | 0.104 [0.050 to 0.171] | 0.132 [0.025 to 0.220] | 0.198 [0.050 to 0.391]

ADVERSE EVENTS:
Arm/Group | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Serious Adverse Events (participants affected / at risk) | 10 | 14 | 10
Other Adverse Events (participants affected / at risk) | 42 | 40 | 35
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Cardio-respiratory arrest (Cardiac disorders) | 1/43 (1) | 1/46 (1) | 0/40 (0)
Angina unstable (Cardiac disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Atrial fibrillation (Cardiac disorders) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Cardiac failure (Cardiac disorders) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Constipation (Gastrointestinal disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Diarrhoea (Gastrointestinal disorders) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Dysphagia (Gastrointestinal disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Chest pain (General disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Bronchiectasis (Infections and infestations) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Cellulitis (Infections and infestations) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Diverticulitis (Infections and infestations) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Gastroenteritis (Infections and infestations) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Urinary tract infection (Infections and infestations) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1/43 (1) | 0/46 (0) | 1/40 (1)
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Cerebrovascular accident (Nervous system disorders) | 2/43 (2) | 0/46 (0) | 1/40 (1)
Grand mal convulsion (Nervous system disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Hemiparesis (Nervous system disorders) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Lethargy (Nervous system disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Parkinson's disease (Nervous system disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Syncope vasovagal (Nervous system disorders) | 0/43 (0) | 1/46 (2) | 0/40 (0)
Confusional state (Psychiatric disorders) | 1/43 (2) | 1/46 (1) | 0/40 (0)
Urinary retention (Renal and urinary disorders) | 1/43 (1) | 0/46 (0) | 1/40 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/43 (0) | 3/46 (5) | 0/40 (0)
Alveolitis fibrosing (Respiratory, thoracic and mediastinal disorders) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Convalescent (Social circumstances) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Suprapubic catheter insertion (Surgical and medical procedures) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Anaemia (Blood and lymphatic system disorders) | 1/43 (1) | 1/46 (1) | 0/40 (0)
Angina pectoris (Cardiac disorders) | 1/43 (1) | 0/46 (0) | 1/40 (1)
Myocardial infarction (Cardiac disorders) | 1/43 (1) | 1/46 (1) | 0/40 (0)
Cardiac failure congestive (Cardiac disorders) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Nausea (Gastrointestinal disorders) | 0/43 (0) | 1/46 (2) | 0/40 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Vomiting (Gastrointestinal disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Asthenia (General disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Catheter related complication (General disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Condition aggravated (General disorders) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Hypersensitivity (Immune system disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Lobar pneumonia (Infections and infestations) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Sepsis (Infections and infestations) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Arthraligia (Musculoskeletal and connective tissue disorders) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Cerebral haemorrhage (Nervous system disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Syncope (Nervous system disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Depression (Psychiatric disorders) | 1/43 (1) | 0/46 (0) | 1/40 (1)
Alcoholism (Psychiatric disorders) | 1/43 (1) | 0/46 (0) | 0/40 (0)
Bladder obstruction (Renal and urinary disorders) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Calculus bladder (Renal and urinary disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
Dysuria (Renal and urinary disorders) | 0/43 (0) | 0/46 (0) | 1/40 (1)
Urine flow decreased (Renal and urinary disorders) | 0/43 (0) | 1/46 (1) | 0/40 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 80/80 + 40 | Degarelix 40/40 + 40 | Degarelix 80 + 20
Anaemia (Blood and lymphatic system disorders) | 2/43 (2) | 3/46 (3) | 2/40 (2)
Atrial fibrillation (Cardiac disorders) | 0/43 (0) | 3/46 (3) | 1/40 (1)
Constipation (Gastrointestinal disorders) | 5/43 (5) | 5/46 (6) | 3/40 (3)
Diarrhoea (Gastrointestinal disorders) | 9/43 (17) | 3/46 (3) | 3/40 (6)
Dyspepsia (Gastrointestinal disorders) | 1/43 (4) | 3/46 (3) | 3/40 (3)
Abdominal distension (Gastrointestinal disorders) | 0/43 (0) | 3/46 (3) | 0/40 (0)
Oedema peripheral (General disorders) | 4/43 (4) | 7/46 (9) | 1/40 (2)
Influenza like illness (General disorders) | 3/43 (8) | 2/46 (2) | 2/40 (2)
Malaise (General disorders) | 3/43 (4) | 0/46 (0) | 0/40 (0)
Lower respiratory tract infection (Infections and infestations) | 6/43 (7) | 6/46 (13) | 3/40 (6)
Urinary tract infection (Infections and infestations) | 7/43 (14) | 3/46 (6) | 4/40 (6)
Nasopharangytis (Infections and infestations) | 3/43 (4) | 5/46 (7) | 2/40 (5)
Injury (Injury, poisoning and procedural complications) | 3/43 (3) | 2/46 (3) | 3/40 (5)
Fall (Injury, poisoning and procedural complications) | 2/43 (2) | 5/46 (5) | 1/40 (1)
Blood cholesterol increased (Investigations) | 4/43 (4) | 5/46 (5) | 2/40 (2)
Gamma-glutamyltransferase increased (Investigations) | 3/43 (4) | 4/46 (5) | 2/40 (2)
Blood alkaline phosphatase increased (Investigations) | 3/43 (3) | 2/46 (3) | 2/40 (2)
Blood creatinine increased (Investigations) | 1/43 (1) | 4/46 (4) | 2/40 (3)
Blood urea increased (Investigations) | 1/43 (1) | 4/46 (4) | 2/40 (3)
Alanine aminotransferase increased (Investigations) | 4/43 (4) | 2/46 (2) | 0/40 (0)
Aspartate aminotransferase increased (Investigations) | 3/43 (3) | 2/46 (2) | 0/40 (0)
Haematocrit decreased (Investigations) | 0/43 (0) | 4/46 (4) | 1/40 (1)
Haemoglobin decreased (Investigations) | 1/43 (1) | 3/46 (4) | 1/40 (1)
Red blood cell count decreased (Investigations) | 0/43 (0) | 4/46 (5) | 1/40 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 3/43 (3) | 1/46 (1) | 0/40 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2/43 (4) | 5/46 (6) | 2/40 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6/43 (6) | 5/46 (5) | 3/40 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2/43 (2) | 1/46 (1) | 4/40 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3/43 (3) | 2/46 (3) | 2/40 (2)
Dizziness (Nervous system disorders) | 2/43 (2) | 4/46 (4) | 3/40 (5)
Headache (Nervous system disorders) | 6/43 (9) | 2/46 (2) | 3/40 (4)
Confusional state (Psychiatric disorders) | 1/43 (2) | 3/46 (4) | 0/40 (0)
Depression (Psychiatric disorders) | 0/43 (0) | 3/46 (4) | 1/40 (1)
Insomnia (Psychiatric disorders) | 3/43 (3) | 3/46 (3) | 1/40 (1)
Nocturia (Renal and urinary disorders) | 4/43 (4) | 4/46 (4) | 1/40 (1)
Dysuria (Renal and urinary disorders) | 3/43 (5) | 2/46 (2) | 3/40 (5)
Pollakiuria (Renal and urinary disorders) | 2/43 (2) | 2/46 (2) | 2/40 (2)
Urinary retention (Renal and urinary disorders) | 0/43 (0) | 3/46 (3) | 0/40 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4/43 (6) | 5/46 (5) | 3/40 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4/43 (4) | 1/46 (1) | 0/40 (0)
Rash (Skin and subcutaneous tissue disorders) | 2/43 (2) | 4/46 (5) | 2/40 (2)
Eczema (Skin and subcutaneous tissue disorders) | 3/43 (4) | 0/46 (0) | 0/40 (0)
Hot flush (Vascular disorders) | 24/43 (25) | 25/46 (25) | 23/40 (27)
Hypertension (Vascular disorders) | 5/43 (6) | 4/46 (5) | 4/40 (4)
Nausea (Gastrointestinal disorders) | 4/43 (5) | 5/46 (6) | 1/40 (1)
Inguinal hernia (Gastrointestinal disorders) | 2/43 (2) | 1/46 (1) | 2/40 (3)
Abdominal pain (Gastrointestinal disorders) | 1/43 (1) | 0/46 (0) | 3/40 (3)
Fatigue (General disorders) | 2/43 (3) | 4/46 (5) | 0/40 (0)
Pyrexia (General disorders) | 3/43 (4) | 1/46 (1) | 0/40 (0)
Suprapubic pain (General disorders) | 0/43 (0) | 0/46 (0) | 2/40 (2)
Cardiac murmur (Investigations) | 0/43 (0) | 1/46 (1) | 2/40 (2)
Weight increased (Investigations) | 0/43 (0) | 0/46 (0) | 2/40 (2)
Gout (Metabolism and nutrition disorders) | 1/43 (1) | 0/46 (0) | 2/40 (2)
Lethargy (Nervous system disorders) | 2/43 (2) | 3/46 (4) | 1/40 (1)
Testicular atrophy (Reproductive system and breast disorders) | 3/43 (3) | 2/46 (2) | 5/40 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3/43 (3) | 0/46 (0) | 0/40 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/43 (0) | 0/46 (0) | 2/40 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3/43 (3) | 3/46 (3) | 1/40 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 3/43 (3) | 0/46 (0) | 0/40 (0)
Flushing (Vascular disorders) | 4/43 (4) | 6/46 (6) | 2/40 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.